CLINICAL TRIAL: NCT05230485
Title: Optimal High CPAP Pressures in Preterm Neonates Post-extubation: A Prospective Randomized Crossover Trial
Brief Title: Optimal High CPAP Pressures in Preterm Neonates Post-extubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Amit Mukerji, Associate Professor, McMaster Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 14289
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Preterm Birth; Mechanical Ventilation Complication; Respiratory Distress Syndrome, Newborn
Keywords: Continuous Positive Airway Pressure; Electrical activity of diaphragm; Continuous distending pressure
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher CPAP (Experimental): CPAP level will be 2 cmH2O higher than pre-extubation measured mean airway pressure
  Interventions: Other: CPAP level
- Equivalent CPAP (Active Comparator): CPAP level will be equal to the pre-extubation measured mean airway pressure
  Interventions: Other: CPAP level

INTERVENTIONS:
Other: CPAP level — The level of continuous distending pressure (or positive end-expiratory pressure) chosen on CPAP

SUMMARY:
Use of continuous positive airway pressure (CPAP) in preterm neonates has traditionally been limited to between 5-8 cmH2O. In recent years, use of CPAP pressures ≥9 cmH2O is becoming more common in neonates with evolving chronic lung disease, in lieu of other non-invasive modes or invasive mechanical ventilation. A particular knowledge gap in the current literature is the choice of the level of pressure level when using High CPAP as a post-extubation support mode. In this study, we will comparatively evaluate the short-term impact of two different high CPAP pressures when used as a post-extubation support mode in preterm neonates.

DETAILED DESCRIPTION:
Background: Use of continuous positive airway pressure (CPAP) in preterm neonates has traditionally been limited to between 5-8 cmH2O. In recent years, use of CPAP pressures ≥9 cmH2O is becoming more common in neonates with evolving chronic lung disease, in lieu of other non-invasive modes or invasive mechanical ventilation. However, there are limited data on the effectiveness and safety of this mode.

A particular knowledge gap in the current literature is the choice of the level of pressure level when using High CPAP as a post-extubation support mode. While it could be argued that the initial High CPAP pressure post-extubation should be somewhat higher than the pre-extubation mean airway pressure (Paw), there remain concerns of potential complications as well as uncertainty around degree of leak and resulting effectiveness. On the other hand, a suboptimal post-extubation High CPAP level may lead to atelectasis and contribute towards extubation failure, potentially prolonging invasive ventilation and associated risks. As such, research towards identification of the optimal High CPAP level post-extubation from high invasive ventilation pressures is warranted.

Objective: To comparatively evaluate the short-term impact of two different high CPAP pressures when used as a post-extubation support mode in preterm neonates.

Hypothesis: We hypothesize that babies extubated from invasive mechanical ventilation with a mean Paw between 9-15 cmH2O will demonstrate better physiological and clinical parameters when using High CPAP+2 cmH2O vs equivalent CPAP levels.

Methods: Design - This will be a prospective, single-centre, randomized cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <29 weeks; chronological age >7 days; post-menstrual age <37 weeks; extubation from invasive ventilation with measured mean airway pressure 9-15 cmH2O

Exclusion Criteria:

* Any congenital or genetic/chromosomal abnormality

Ages: 7 Days to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Peak Edi | 60 min following each CPAP level - assessed over 10 min
  The peak electrical diaphragmatic activity - a surrogate for work of breathing to generate tidal volume

SECONDARY OUTCOMES:
Minimum EDi | 60 min following each CPAP level - assessed over 10 min
  The minimum eelectrical diaphragmatic activity - a surrogate for work of breathing to maintain functional residual capacity
Regional cerebral perfusion | 60 min following each CPAP level - assessed over 10 min
  The cerebral tissue extraction of oxygen - determined by near infra-red spectroscopy
Pressure level - Ventilator | 60 min following each CPAP level - assessed over 10 min
  Pressure level as measured by the ventilator
Pressure level - Interface | 60 min following each CPAP level - assessed over 10 min
  Pressure level at measured at the nasal interface used to deliver CPAP
Work of breathing score | Over entire duration (70 min) at each CPAP level, assessed every 10 min
  Using Silverman Scoring
Heart Rate | Over entire duration (70 min) at each CPAP level, assessed every 10 min
  From cardiorespiratory monitoring
Respiratory Rate | Over entire duration (70 min) at each CPAP level, assessed every 10 min
  From cardiorespiratory monitoring
Transcutaneous CO2 level | Over entire duration (70 min) at each CPAP level, assessed every 10 min
  From bedside transcutaneous CO2 monitoring
FiO2 level | Over entire duration (70 min) at each CPAP level, assessed every 10 min
  Fractional inspired oxygen level, as determined by clinical and inputted into ventilator
Number of bradycardic episodes <80 bpm | Over entire duration (70 min) at each CPAP level
  as above
Proportion of duration with SpO2 <90% | Over entire duration (70 min) at each CPAP level
  duration of time where the patient's SpO2 is less than 90%

CONTACTS AND LOCATIONS:
Overall Officials: Amit Mukerji, MD, Principal Investigator — Associate Professor
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No